CLINICAL TRIAL: NCT04233320
Title: Efficacy and Safety of Silicone Cream Containing Allium Cepa Extract in Post-cesarean Surgical Scars Treatment
Brief Title: Efficacy and Safety of Silicone Cream Containing Allium Cepa Extract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 547/62
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Cicatrix
Keywords: Scar; Allium Cepa; post-cesarean
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- silicone cream containing Allium Cepa extract (Experimental): Silicone cream containing Allium Cepa extract will be applied on half of post-cesarean surgical scars 2 times per day for 3 months.
  Interventions: Device: silicone cream containing Allium Cepa extract
- commercial scar gel (Active Comparator): Commercial scar gel will be applied on half of post-cesarean surgical scars 2 times per day for 3 months.
  Interventions: Device: Commercial scar gel

INTERVENTIONS:
Device: silicone cream containing Allium Cepa extract — silicone cream containing Allium Cepa extract contains 10% of Allium cepa bulb extract.
  Arms: silicone cream containing Allium Cepa extract
Device: Commercial scar gel — Commercial scar gel is a topical silicone gel. It contains cyclic and polymeric siloxanes and Vitamin C ester.
  Arms: commercial scar gel

SUMMARY:
The objectives of this study were to evaluate efficacy and safety of silicone cream containing Allium Cepa extract in post-cesarean surgical scars treatment. Post-cesarean surgical scars were equally seperated into 2 parts (left part and right part). Silicone cream containing Allium Cepa extract or commercial scar gel was ramdomly assigned to apply on left part or right part of the scar. They will be applied 2 times per day (morning and evening) for 3 months. Patient and Observer Scar Assessment Scale (POSAS) , Vancouver scar scale (VSS), melanin index, and erythema index (using cutometer) were used for scar evaluation at 0, 1,2,and 3 months. Moreover, adverse effects were also observed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Have Post-Cesarean Surgical Scars at least 1 month
* REEDA scale = 0 score
* Able to read and write Thai
* Able to follow the research plan
* Able to meet all the researchers throughout the period of participation in the project

Exclusion Criteria:

* Apply other topical application at the post-cesarean surgical scars within 2 weeks before participating in the study and during the study
* There is radiation in the area of the post-cesarean surgical scars
* Chronic skin diseases such as psoriasis, chronic dermatitis, allergies
* Immune deficient or use immunosuppressants within 2 weeks before participating in the study and during the study
* Have a history of silicone allergy or onion extract

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale | 3 months
  The range of score is 1 to 10. Noraml skin will be recorded as scale 1. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Vancouver scar scale | 3 months
  The range of score is 0 to 10. Higher scores mean a worse outcome.
Melanin index | 3 months
  Melanin index will be evaluated using cutometer.
Erythema index | 3 months
  Erythema index will be evaluated using cutometer.
Adverse effect | 3 months
  Adverse effect will be observed in term of erythema, edema, papules, vesicles, and bullae. The range of erythema score is 0 to 3. The range of edema score is 0 to 4. Higher scores mean a worse outcome. Papules, vesicles, and bullae will be recorded as apperance or clear.

IPD SHARING:
Plan to Share IPD: No